CLINICAL TRIAL: NCT06495437
Title: Preliminary Safety and Efficacy Study of Extracellular Vesicle Infusion in the Intervention of Age-related Phenotypes With Impaired Glucose Tolerance.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BEAUTECH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91469002MA5RCDY83W
Record Dates: First submitted 2024-06-13; First posted 2024-07-10 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Impaired Glucose Tolerance
Keywords: Extracellular Vesicle; Aging; Human Mesenchymal Stem Cells; impaired glucose tolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm study (Experimental): Subjects who met the inclusion criteria were intravenously infused with 100ml extracellular vesicles derived from umbilical cord mesenchymal stem cells, at a rate of 1-1.5 hours
  Interventions: Biological: Intravenous infusion of extracellular vesicle preparation derived from Wharton's jelly mesenchymal stem cells.

INTERVENTIONS:
Biological: Intravenous infusion of extracellular vesicle preparation derived from Wharton's jelly mesenchymal stem cells. — The trial protocol includes a 3-week screening period and a 12-week study period after enrollment. The specific trial protocol is detailed in the figure above. Cell-derived extracellular vesicle formulation will be administered at week 0, with central visits conducted during the administration period. Central visits will also be conducted at weeks 1, 4, and 12 post-administration, with a phone visit at week 8. The entire study will last for 12 weeks. Following the final follow-up visit, further observation of the intervention's effects and safety will continue for an additional 3 months. During this 3-month period, there will be no artificial intervention or restriction on the medication and biological methods for the participants in each group.

SUMMARY:
The objective of this exploratory study was to evaluate the initial safety of human mesenchymal stem cell-derived extracellular vesicle infusion in an age-related phenotype with impaired glucose tolerance

ELIGIBILITY:
Inclusion Criteria:

1. The subjects are between 35 and 65 years old (inclusive), regardless of gender;
2. The subject's body mass index (BMI) is between 20kg/m2 and 30 kg/m2;
3. The subjects were assessed by the clinical expert group as having abnormal glucose tolerance (PPG 7.8-11.0mmol/L 2h postprandial);
4. Subjects voluntarily participate in this clinical study and sign a written informed consent.

Exclusion Criteria:

1. The subject has a severe allergy or is allergic to any component used in cell culture;
2. The subject has used or is using drugs that affect glucose metabolism (such as glucocorticoids, tricyclic antidepressants, etc.) within 1 month;
3. The subjects have chronic diseases such as diabetes and hypertension (very high-risk group) which have not been effectively controlled after treatment;
4. Subjects with severe cardiovascular and cerebrovascular diseases: patients with a history of decompensated cardiac insufficiency (NYHA grade Ⅲ or Ⅳ), myocardial infarction or cerebral infarction, or cerebral hemorrhage within 6 months before screening;
5. The subjects had abnormal liver function (ALT and/or AST≥ 2.5 times the upper limit of normal), significant abnormal renal function, male serum creatinine ≥1.5mg/dl, female serum creatinine ≥1.4mg/dl; 6, the subject's HIV antibody, hepatitis B surface antigen, hepatitis C antibody, syphilis test positive, hepatitis B virus DNA quantitative > the upper limit of normal test unit;

7. Subjects with other serious systemic diseases affecting the study, including malignant tumors, nervous central system, blood system, digestive system, endocrine system, respiratory system, infectious diseases, etc.; (8) Drug or alcohol abuse (subjects who consumed >2 alcoholic beverages per day or >14 alcoholic beverages per week (one alcoholic beverage is defined as 150ml of wine, 350ml of beer, or 50ml of 80% (40 proof) spirits); Or drug abusers; 9. Pregnant and lactating women; Have a pregnancy plan in the next 2 years (including the spouse's pregnancy plan); Refusal to use effective contraception; 10. Exclude intracranial lesions and early lung tumors; 11. Used stem cell (exosome) therapy or participated in stem cell (exosome) clinical researchers 3 months before screening; Clinical investigators who have participated in drugs within 3 months before screening; 12. High risk groups with Padua score ≥4 or Caprini score ≥5; 13. The subject has a history of major surgery within the past six months or is expected to have surgery within six months; 14. There are other conditions that the researcher considers inappropriate to participate in this clinical study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
safety evaluation | 0-12 weeks
  Incidence of adverse events from baseline to the end of 12 weeks. The frequency and frequency of adverse events (including injection site reactions) were analyzed. The number of cases and cases of adverse events, adverse reactions, AES leading to fall off, SAE, aes of different severity, AES leading to death were calculated respectively, and a detailed list was provided. The incidence rate was calculated using the number of people in each safety dataset as the denominator, and if necessary, Chi-square test or Fisher exact probability method was used for inter-group comparison.

SECONDARY OUTCOMES:
Effectiveness evaluation | 0-12 weeks
  glycated hemoglobin -1
Effectiveness evaluation | 0-12 weeks
  endocrine hormones (gonadal hexa, DHEA, IGF-1)
Effectiveness evaluation | 0-12 weeks
  blood glucose level
Effectiveness evaluation | 0-12 weeks
  insulin secretion index
Effectiveness evaluation | 0-12 weeks
  HOMA-β indexes
Effectiveness evaluation | 0-12 weeks
  HOMA-IR indexes